CLINICAL TRIAL: NCT07392528
Title: A Clinical Study Evaluating the Safety and Preliminary Efficacy of Universal Allogeneic CAR T-cell Therapy Targeting CD19 and BCMA（QT-019C） in Patients With Relapsed / Refractory Neurological Autoimmune Diseases
Brief Title: Universal Chimeric Antigen Receptor T-Cell （UCAR T-cell） Therapy Targeting CD19/ BCMA（QT-019C） in Patients With r/ r Neurological Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Jialing Wu, Principal Investigator, Tianjin Huanhu Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH-HH-03
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neuromyelitis Optica Spectrum Disorders; Multiple Sclerosis; Myasthenia Gravis
Keywords: Universal Allogeneic CAR T-cells; QT-019C
MeSH Terms: conditions — Neuromyelitis Optica; Multiple Sclerosis; Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QT-019C (Experimental): Universal allogeneic CD19/BCMA CAR T-cells
  Interventions: Drug: QT-019C

INTERVENTIONS:
Drug: QT-019C — Universal allogeneic anti-CD19/BCMA CAR T-cells

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 15 participants with relapsed or refractory Neurological Autoimmune Diseases. This study aims to evaluate the safety and efficacy of the treatment with universal CD19/BCMA CAR T-cells（QT-019C）.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal CD19/BCMA CAR T-cells（QT-019C） in Relapsed or Refractory Neurological Autoimmune Diseases.Study intervention consists of a single infusion of universal CAR T-cells administered intravenously after a lymphodepleting therapy regimen of cyclophosphamide.Interim analysis will be performed when participants finish the visit 90 days after CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Subjects with relapsed or refractory neurological autoimmune diseases, Including neuromyelitis optica spectrum disorders(NMOSD), myasthenia gravis(MG), multiple sclerosis(MS)，Autoimmune encephalitis(AE) and chronic inflammatory demyelinating Polyradiculoneuropathy(CIDP).
* Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically approved contraception or abstinence during the study treatment period and for at least 6 months after the end of the study treatment; Female subjects of childbearing potential must have a negative Human chorionic gonadotropin (HCG) test within 7 days before study enrollment and not be lactating.
* Willing to participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Subjects with a history of severe drug allergies or allergic tendencies.
* History of malignancy within five years. The following conditions are excluded: non-melanoma skin cancer, stage I tumors that have a low recurrence probability after complete resection, clinically localized prostate cancer after treatment, cervical carcinoma in situ confirmed by biopsy or squamous intraepithelial lesion shown on smear, stable papillary thyroid carcinoma or follicular thyroid carcinoma.
* Subjects with insufficient cardiac function.
* Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA >the upper limit of detection; subjects positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; individuals positive for human immunodeficiency virus (HIV) antibody; individuals positive for syphilis testing.
* Pregnant women or women planning to conceive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The number and severity of dose-limiting toxicity (DLT) events | Within 28 Days After QT-019C Infusion
  DLT will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, and the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells.
The total number, incidence, and severity of AEs | Up to 90 days After QT-019C Infusion

SECONDARY OUTCOMES:
NMOSD、MS: Expanded Disability Status Scale (EDSS) score | Up to 24 Months After QT-019C Infusion
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS is a scale for assessing neurologic impairment in multiple sclerosis (MS). It consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death from MS). A negative change from baseline indicates improvement. A participant was considered to have a worsening in overall EDSS score of at least 2 if baseline EDSS score was 0, or at least 1 point if baseline EDSS score is 1 to 5, or at least 0.5 point if baseline EDSS score is 5.5 or more.
NMOSD、MS: Modified Rankin Scale | Up to 24 Months After QT-019C Infusion
  Modified Rankin Scale (mRS) is a profoundly valid and reliable measure of disability and is broadly utilized for assessing stroke outcomes and degree of disability. We characterized a favorable outcome as mRS ranging from zero up to two, while unfavorable outcome ranging for 3 up to 6.
MG: Quantitative Myasthenia Gravis Score (QMG) | Up to 24 Months After QT-019C Infusion
  The QMG score is a 13-item scale used to quantify disease severity in myasthenia gravis. The scale measures ocular, bulbar, respiratory, and limb function, grading each finding, and ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits).
MG: Myasthenia Gravis Activities if Daily Living (MG-ADL) Score | Up to 24 Months After QT-019C Infusion
  The MG-ADL is an eight-question survey of symptom severity, with each response graded from 0 (normal) to 3 (most severe). Two questions concern ocular, three oropharyngeal, one respiratory, and two extremity functions. Cumulative MG-ADL scores range from 0 to 24
CIDP: Inflammatory Neuropathy Cause and Treatment (INCAT) Score | Up to 24 Months After QT-019C Infusion
  The INCAT score comprises two parts, the arm score and the leg score. Based on a patient's level of impairment in their arms and legs, each part is scored between 0 and 5 points, resulting in an INCAT total score between 0 and 10.
AE: Change in CASE | Up to 24 Months After QT-019C Infusion
  The changes of Clinical Assessment Scale in Autoimmune Encephalitis (CASE) score from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, China